CLINICAL TRIAL: NCT04210440
Title: Core Decompression With Bone Chips Allograft Adjuvanted by Fibrin Platelet Rich-plasma (PRP) and Concentrated Autologous Mesenchymal Stromal Cells (MSCS): Results in Avascular Necrosis of Femoral Head (AVN) After 2 Years Minimum Follow-up
Brief Title: The Treatment of Initial Stage of Hip Osteonecrosis: the Core Decompression
Acronym: NEC15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dante Dallari, MD (Other)
Responsible Party: Sponsor-Investigator, Dante Dallari, MD, MD, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0029170
Record Dates: First submitted 2019-12-21; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Hip Necrosis; Hip Injuries
Keywords: hip avascular necrosis; hip conservative surgery
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip avascular necrosis (Experimental): patients affected by avascular necrosis of the Hip classified by Japanese Investigation Committee criteria
  Interventions: Procedure: Core decompression procedure

INTERVENTIONS:
Procedure: Core decompression procedure — Core Decompression with Bone Chips Allograft adjuvanted by Fibrin Platelet Rich-plasma (PRP) and Concentrated Autologous Mesenchymal Stromal Cells (MSCS), isolated from Bone Marrow

SUMMARY:
This retrospective study evaluates 52 cases of avascular necrosis of femoral head (AVN) treated by core decompression, bone chips allograft, fibrin platelet rich-plasma (PRF) and concentrated autologous mesenchymal stromal cells (MSCs).

DETAILED DESCRIPTION:
We report 52 cases of avascular necrosis of the hip (AVN), operated by decompression of the necrotic area with bone chips allograft, adjuvanted by concentrated autologous mesenchymal stromal cells (MSCs) and fibrin platelet rich-plasma (PRP).

The patients were followed-up at 6 weeks, 3 months, 6 months, 12 months, 24 months and then every year. Each time a clinical evaluation by Harris Hip Score (HHS) was carried out by the same orthopedic surgeon. Radiological controls (pelvis and hip affected) were performed at 6 weeks, 3 months, 6 months, 12 months, 24 months and then every year.

The primary outcome evaluated was the avoiding or delaying of total hip replacement (THR), while the secondary outcomes were the assessment of any change in clinical performance as measured by Harris Hip Score

ELIGIBILITY:
Inclusion Criteria:

- hip avascular necrosis

Exclusion Criteria:

* protrusio acetabuli
* concentric femoral head migration;
* presence of extensive surgery of the reference joint (osteotomies around the hip, open or arthroscopic osteochondroplasty for femoral-acetabular impingement)
* presence of excessive deformity (acetabular or femoral head dysplasia; collapse deformity and deformed femoral head sequelae of Perthes);
* concomitant rheumatic diseases;
* bone tumors

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2003-03-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Avoiding arthroplasty | 24 months after surgery
  The primary outcome evaluated was the avoiding or delaying of total hip replacement (THR)

SECONDARY OUTCOMES:
Harris Hip Score | 6 weeks after surgery
  The collection of functional outcomes score HHS at 6 weeks. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
Harris Hip Score | 3 months after surgery
  The collection of functional outcomes score HHS at 3 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results
Harris Hip Score | 6 months after surgery
  The collection of functional outcomes score HHS at 6 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.
Harris Hip Score | 12 months after surgery
  The collection of functional outcomes score HHS at 12 month after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 as poor result; 70-80 as fair, 80-90 as good, and 90-100 as excellent results.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzli, Bologna, Italy